CLINICAL TRIAL: NCT05013996
Title: Impact d'un Bilan Clinique structuré (MIDSA), de sa Restitution et de l'Accompagnement au Changement Sur l'Engagement Dans le Soin (évalué Par l'échelle URICA) d'Auteurs d'Infraction à caractère Sexuel : Essai contrôlé randomisé Multicentrique en Ouvert
Brief Title: Impact of a Structured Clinical Assessment MIDSA, Its Feedback and Support for Change on Commitment to Care of Perpetrators of Sexual Offenses
Acronym: EV-AICS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 10 patients out of 152 expected over 3 years of inclusion. There are many reasons for this failure (staff recruitment, duration of MIDSA..).
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EV-AICS (DR190059); 2020-A02628-31 (Registry Identifier: Id-RCB-ANSM-France); DR190059 (Other: Sponsor Reg n°)
Record Dates: First submitted 2021-06-03; First posted 2021-08-20 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Offense, Sex
Keywords: sexual offenders;MIDSA
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Intervention Model Description: open label multicenter randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized to the experimental (MIDSA groupe) will be treated according to the usual methods of each of the centers (CMP / CRIAVS / private practitioners, etc.) completed with the Multidimensional Inventory of Development, Sex, and Aggression-MIDSA groupe Multidimensional Inventory of Development, Sex, and Aggression-inventory tool.
  Interventions: Behavioral: MIDSA
- Control (Active Comparator): Patients randomized to the control group will be treated according to the usual methods of each of the participating centers (CMP / CRIAVS / private practitioners, etc.).
  Interventions: Behavioral: Usual methods of evaluation

INTERVENTIONS:
Behavioral: MIDSA — Multidimensional Inventory of Development, Sex, and Aggression
  Arms: Intervention
Behavioral: Usual methods of evaluation — Usual methods of evaluation of each of the participating centers (CMP / CRIAVS / private practitioners, etc.).
  Arms: Control

SUMMARY:
Evaluate the effectiveness of an intervention including the clinical assessment carried out with the (Multidimensional Inventory of Development, Sex, and Aggression) MIDSA and the review of the results with the professional in charge of the subject on the adherence and commitment to the care of the sexual offenders.

DETAILED DESCRIPTION:
The intervention of MIDSA (Multidimensional Inventory of Development, Sex, and Aggression), a multidimensional investigation tool for issues related to sexuality and violence, could be prove very useful by providing AICS patients as well as the professionals who take care of them with a complete clinical assessment which enlightens the patient on his psychopathological functioning and / or his disorders, and which guides the care through the axes of intervention to be implemented in response to the criminological and non-criminological needs of the patient. This should allow the latter a better awareness (awareness) of his difficulties in the relationship with the other, facilitate his adherence to care, obtain a better commitment on his part in the process of change and consequently, bring him change their lifestyle and gradually adopt proactive attitudes and behavior that ultimately reduce the risk of recidivism of sexual and general violence. However, recourse to MIDSA as a "change operator" in a patient's trajectory is only possible if it is accompanied by a resumption of his clinical assessment by a professional who supports the change process by strengthening his motivation to change their criminal behavior.

ELIGIBILITY:
Inclusion Criteria:

* Adult male patients
* Express written consent of the participant after receiving the study information
* Subject making contact or being taken in charge by a psychiatric service (even an addictology service or by liberal practitioners in connection with psychiatry), a CRIAVS or a care unit dedicated to the care of perpetrators of a sexual offense (AICS) ;
* For a problem of sexual violence such as sexual harassment, assault and rape of adult women (including marital rape), incest, pedophilic or hebephilic acts, sexual sadism, exhibition, voyeurism, frotteurism, use and possession of child pornography or addiction sexual.

  * Affiliated to a social security scheme

Exclusion Criteria:

* Maximum stage (maintenance phase) listed on the URICA scale
* Poor understanding of the French language;
* Patient imprisoned, under legal protection, under guardianship or curatorship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult male patients
Enrollment: 10 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Change in behavior | up to 6 months
  Change in behavior (awareness of its difficulties, commitment to care, motivation to abandon the previous lifestyle, etc.) and with reference to the transtheoretical model of stage change, it will be measured using the University of Rhode Island Change Assessment (URICA) by the rate of patients with a stage of change at Month 6 higher than that observed at D0

SECONDARY OUTCOMES:
Assessment of the risk for sexual violence (RSVP) | up to 1 year
  The risk assessment for sexual violence will be performed by the Risk for Sexual Violence Protocol (RSVP; Hart et al., 2003);cut-off score: 0-44 (lowrisk); score: 45-132 moderate to high risk
Assessment of the risk of violence (in general) and the risk factors of the sexual offenders | up to 1 year
  The assessment of the risk of violence (in general) and the risk factors of the sexual offenders will be carried out from the Level of Service Inventory / Case Management Inventory (LS / CMI; Andrews , Bonta, & Wormith, 2000; Guay, 2008);
Assessment of the multidimensional self-esteem assessment (SEI) | up to 1 year
  The multidimensional self-esteem assessment will be carried out by the Self-Esteem Inventory (SEI; Coopersmith, 1981) with 4 dimensions: general, social, family and professional self-esteem;
Quality of life assessment | up to 1 year
  The quality of life assessment will be carried out by the World Health Organization Quality Of Life (WHOQOL-brief); Leplege, Reveillere, Ecosse, Caria, & Riviere, 2000; The WHOQOL Group, 1998) around four dimensions: physical health, psychological health, social relations and the environment.
Assessment of social desirability will be carried out by the MCSDS | up to 1 year
  The assessment of social desirability will be carried out by the Marlow-Crowne Social Desirability Scale (MCSDS) through its brief version of 20 items
Assessment of Risk factors and protective factors against violence | up to 1 year
  Risk factors and protective factors against violence are assessed through a semi-structured interview (for assessment of Risk for Sexual Violence Protocol (RSVP), Level of Service Inventory/Case Management Inventory (LS / CMI) and Structured Assessment of Protective Factors (SAPROF))

CONTACTS AND LOCATIONS:
Overall Officials: Robert COURTOIS, MD-PhD, Study Director — University Hospital of TOURS
Locations (5):
- France (5):
  - CHRU Lille - URSAVS Lille, Lille
  - CH LE Vinatier - Service de Psychiatrie Légale, Lyon
  - CHU Montpellier Lapeyronie - CRIAVS Languedoc-Roussillon, Montpellier
  - CHU Poitiers Henri Laborit - CRIAVS - CMP Espace Vienne - SMPR, Poitiers
  - CHRU Tours - UC3P, Tours

IPD SHARING:
Plan to Share IPD: No